CLINICAL TRIAL: NCT00771264
Title: Study of Urgent PC Versus Sham Effectiveness in Treatment of Overactive Bladder Symptoms
Acronym: SUmiT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uroplasty, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UPC082008
Record Dates: First submitted 2008-10-09; First posted 2008-10-13 (Estimated); Results first posted 2010-09-21 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Urgent PC (Active Comparator)
  Interventions: Device: Urgent PC Neuromodulation System
- Sham / Placebo (No Intervention)

INTERVENTIONS:
Device: Urgent PC Neuromodulation System — The Urgent PC Neuromodulation System is a minimally invasive neuromodulation system designed to deliver retrograde access to the sacral nerve through percutaneous electrical stimulation of the tibial nerve. The method of treatment is referred to as Percutaneous Tibial Nerve Stimulation (PTNS).
  Arms: Urgent PC

SUMMARY:
The purpose of this study is to demonstrate superiority of percutaneous posterior tibial nerve stimulation (PTNS) therapy compared to sham therapy for the treatment of patients with overall bladder (OAB) symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Women and men >18 years of age
* A score of > 4 on the OAB-q short form for urgency (question 1)
* Average urinary frequency > 10 times in one 24 hour day based on a 3-day voiding diary
* Self-reported bladder symptoms present > 3 months
* Self-reported failed conservative care (i.e., dietary restriction, fluid restriction, bladder training, behavioral modification, pelvic muscle training, biofeedback, etc.)
* Off all antimuscarinics for at least 2 weeks prior to enrollment
* Capable of giving informed consent
* Ambulatory and able to use a toilet independently, without difficulty
* Capable and willing to follow all study-related procedures

Exclusion Criteria:

* Pregnant as confirmed by urine pregnancy test, or plans to become pregnant during the study period
* Neurogenic bladder
* Botox use in bladder or pelvic floor muscles in the past year
* Pacemakers or implantable defibrillators
* Primary complaint of stress urinary incontinence
* Current urinary tract infection (UTI)
* Current vaginal infection
* Current use of InterStim
* Current use of Bion
* Current use of TENS in the pelvic region, back or legs
* Previously been treated with PTNS
* Use of investigational drug/device therapy within the past 4 weeks
* Participating or have participated within the past 4 weeks in any clinical investigation involving or impacting gynecologic, urinary or renal function
* Deemed unsuitable for enrollment in study by the investigators based on subjects' history or physical examination (including bleeding disorders or anticoagulant medications, and peripheral neuropathy)
* Subjects with nerve damage that would impact either percutaneous tibial nerve or pelvic floor function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Gregory L. Davis, M.D., FACOG, Inc., Chico, California
  - Greenwich Urological Associates, P.C., Greenwich, Connecticut
  - Specialists in Urology, Naples, Florida
  - Mercy Health Partners at the Lakes, Muskegon, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Grand Rapids Women's Health DBA Female Pelvic Medicine & Urogynecology Institue of Michigan, Grand Rapids, Minnesota
  - Uroplasty, Inc, Minnetonka, Minnesota
  - Beaumont Hospital, Royal Oak, Minnesota
  - Urology Health Center, PC, Fremont, Nebraska
  - Capital Region Urological Surgeons, PLLC, Albany, New York
  - Central Missouri Women's Healthcare, LLC, White Plains, New York
  - Alliance Urology Specialists, Greensboro, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Virginia Urology, Richmond, Virginia
  - Athena Urology, Issaquah, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by investigator sites with limited advertising
Period: Overall Study
Arm/Group | Urgent PC | Sham / Placebo
Started | 110 | 110
Completed | 103 | 105
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Urgent PC | Sham / Placebo | Total
Number analyzed (Participants) | 110 | 110 | 220
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 64 | 118
  >=65 years | 56 | 46 | 102
Age Continuous [Mean (Standard Deviation); unit: years] | 62.5 (14.6) | 60.2 (15.2) | 61.3 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 88 | 174
  Male | 24 | 22 | 46
Region of Enrollment [Number; unit: participants]
  United States | 110 | 110 | 220

OUTCOME MEASURES:

1. Primary Outcome: The Global Response Assessment (GRA) for Overall Bladder Symptoms to Compare the Proportion of Subjects Reporting "Moderately" or "Markedly Improved" Responses on the GRA After 12 Interventions of Randomized Therapy, in an Intent to Treat Analysis.
Description: A responder was defined as reporting bladder symptoms as moderately or markedly improved on a 7-level GRA at week 13 after completing 12, 30-minute, consecutive weekly intervention sessions.
Time Frame: 13 weeks
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Urgent PC | Sham / Placebo
Number analyzed (Participants) | 110 | 110
participants | 60 | 23
Statistical Analysis 1: Comparison: Urgent PC vs Sham / Placebo; Mean values were analyzed for significant change using a 2-sided paired t test and proportions were analyzed using chi-square methodology. Median values were analyzed using a Wilcoxon signed rank test with p<0.05 considered statistically significant. A sample size estimate of 214 subjects, 107 per arm, was calculated using a 2-sided Fisher's exact binomial test based on an estimated 60% responder rate in the PTNS group and a 40% in the sham group with a 5% significance level and 80% power; Test type: Superiority or Other; p = 0.05, t-test, 2 sided — P-values <0.05 were considered statistically significant; Mean values were analyzed for significant change using a 2-sided paired t-test and proportions were analyzed using chi-square methodology

ADVERSE EVENTS:
Arm/Group | Urgent PC | Sham / Placebo
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/110
Other Adverse Events (participants affected / at risk) | 6/110 | 0/110
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Urgent PC (N=110) | Sham / Placebo (N=110)
ankle bruising (Surgical and medical procedures) | 1 (1) | 0 (0)
discomfort at needle site (Surgical and medical procedures) | 2 (2) | 0 (0)
bleeding at needle site (Surgical and medical procedures) | 3 (5) | 0 (0)
tingling in leg (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No